CLINICAL TRIAL: NCT01050725
Title: Investigating Proteomic Biomarkers of Radiation Therapy Outcome: A Pilot Study
Brief Title: Pilot Study of Biomarkers for Radiation Therapy
Status: Suspended | Type: Observational
Why Stopped: On hold: pending grant funding for further enrollment
Sponsor: Benaroya Research Institute (Other)
Collaborators: Virginia Mason Hospital/Medical Center (Other); Fred Hutchinson Cancer Center (Other)
Responsible Party: Kas Badiozamani, Virginia mason Medical Center
Other Study IDs: IRB09016
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Cancer
Keywords: proteome; biomarkers; radiotherapy; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: whole blood samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Radiation therapy patients: Individuals receiving radiation therapy as definitive or neo-adjuvant therapy for selected malignancies, including head and neck, lung, esophageal, rectal cervical and prostate cancers.

SUMMARY:
The purpose of this study is to determine whether specific assays of DNA damage repair proteins can be used in patients undergoing radiation therapy. The ultimate goal of this research is to develop clinically useful biomarkers from blood samples that could be used to customize radiation treatment for individuals, leading to reduced side effects and improved outcomes.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years of age with primary lung, esophageal or rectal cancer receiving neo-adjuvant chemoradiotherapy before planned resection
* patients with clinically localized prostate cancer receiving definitive radiation therapy with external beam treatment. brachytherapy as a boost and/or hormonal therapy are allowed.
* patients with head and neck, lung, esophageal or cervical cancer who will receive definitive radiotherapy

Exclusion Criteria:

* prior history of chemotherapy given within 6 months before enrollment.
* prior radiotherapy or radionuclide treatment and/or brachytherapy within 6 months prior to enrollment.
* unwillingness to comply with tests, protocol, or informed consent.
* concurrent enrollment on any protocol that would require non-compliance with treatment procedures.
* chemotherapy required within 2 hours following first dose of XRT.
* PET scan done within 48 hours of first blood draw.
* nuclear medicine exposure within 4 days prior to first draw.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing radiation for selected malignancies, including head and neck, lung, esophageal, rectal, cervical and prostate cancers.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-11; Primary Completion 2013-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kas R Badiozamani, MD, Principal Investigator — Virginia Mason Hospital/Medical Center
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States